CLINICAL TRIAL: NCT06359847
Title: A Multicenter, Phase II Clinical Trial to Evaluate the Efficacy and Safety of ST-1898 Tablets in Patients With Locally Advanced or Metastatic RAIR-DTC After Failure of at Least First-line TKI Systemic Therapy
Brief Title: Study of ST-1898 in Locally Advanced or Metastatic Radioiodine-Refractory Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Scitech-Mq Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-1898-202
Record Dates: First submitted 2024-01-03; First posted 2024-04-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Differentiated Thyroid Carcinoma
Keywords: ST-1898，Differentiated Thyroid Cancer
MeSH Terms: interventions — 3-(3'-adamantan-1-yl-4'-methoxybiphenyl-4-yl)-2-propenoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ST-1898 (Experimental): ST-1898 tablet is administered orally at 180 mg once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21), until disease progression or intolerable toxicity.
  Interventions: Drug: ST-1898 tablets

INTERVENTIONS:
Drug: ST-1898 tablets — Tablets: 5 mg and 40 mg

SUMMARY:
ST-1898, a multi-targeted tyrosine kinase inhibitor, has demonstrated strong inhibitory activity for VEGFR2, c-MET, AXL, PDGFRA, RET, KIT, etc. The primary purpose of this study is to evaluate the efficacy of ST-1898 tablets in patients with locally advanced or metastatic RAIR-DTC after failure of at least first-line TKI systemic therapy. All subjects will receive ST-1898 180 mg orally once daily until disease progression or intolerable toxicity.

ELIGIBILITY:
Eligibility Minimum Age: 18 Years

Maximum Age:

Sex: All

Gender Based:

Accepts Healthy Volunteers: No

Criteria: Inclusion Criteria:

1. Age >= 18 years
2. Life expectancy of twelve weeks or more
3. Histologically or cytologically confirmed locally advanced or metastatic DTC that cannot be removed by surgery or radiotherapy, including papillary thyroid cancer, follicular thyroid cancer, hurthle cell thyroid cancer or poorly differentiated thyroid cancer.
4. At least one measurable lesion according to RECIST 1.1
5. Radioiodine-refractory (RAI-refractory) differentiated thyroid cancer can be diagnosed when any of the following criteria are met under thyroid-stimulating hormone (TSH) stimulation (>30 mU/L) in the absence of exogenous iodine interference:

   * Negative uptake in one or more measurable lesions after receiving I-131 treatment or scanning
   * One or more measurable lesions that has progressed as per RECIST 1.1 within 14 months of 131I therapy（3.7~7.4 GBq or100~200 mCi）,despite demonstration of radioiodine avidity at the time of that treatment by pre- or post-treatment scanning.
   * Cumulative activity of 131I of > 22 GBq or 600 mCi, with the last dose administered at least 6 months prior to study entry
6. Subjects with DTC who failed with or was intolerant to at least one prior tyrosine kinase inhibitor (TKI) therapy. If prior treatment with VEGFR-TKI, no more than two VEGFR-TKIs were allowed.
7. Recommendation of subject offering archived tissue sample or previous biomarker of MET test report. If archived tumor sample is not available, a fresh biopsy is optional, which need to be taken from needle biopsy or core needle biopsy (fine needle biopsy not allowed). Subjects who cannot provide tissue samples or test reports may still be eligible to participate if the investigator determines a potential clinical benefit from ST-1898 therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. TSH-suppression therapy is well tolerated with thyroid stimulating hormone (TSH) < 0.5 mU/L;
10. The patient has adequate organ and bone marrow function as follows:

    * Adequate bone marrow function (without transfusion or colony stimulating factor support within 2 weeks): hemoglobin ≥ 90 g/L, absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L and platelets ≥ 100 × 10^9/L;
    * Adequate liver function: Bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 × ULN (≤ 5 × ULN if participant has liver metastases);
    * Adequate renal function: Serum creatinine ≤1.5 ×ULN or creatinine clearance≥50 mL/min per the Cockcroft-Gault formula;
    * Adequate blood coagulation function: International Normalized Ratio (INR) ≤ 1.5 and Activated partial thromboplastin time (APTT) ≤1.5 ULN（except for the prophylactic use of anticoagulants）
    * Adequate cardiac function: Left ventricular ejection fraction (LVEF) ≥50%;
    * Participants having≤ 1 + proteinuria or ≥2+ proteinuria with urine protein < 1 g/24 hour.
11. Ability to understand and the willingness to sign a written informed consent document. The results of routine examination during the corresponding window period before screening are acceptable.
12. Women with child-bearing potential and men must agree to use adequate contraception (e.g., hormonal contraceptives, male or female condom, or abstinence) during the course of the study and for at least 3 months following the last dose of study drug. Women with childbearing potential must have a negative serum pregnancy test within 7 days before first study treatment.

Exclusion Criteria:

1. Other histological subtypes of thyroid cancers excluding DTC (such as Anaplastic Thyroid Carcinoma and Medullary Thyroid Carcinoma).
2. Known hypersensitivity to any component of ST-1898 tablets.
3. Participants who have received any antitumor treatment within 4 weeks or 5 half-lives of the agent (contingent on the shorter time) prior to the first dose of study drug.
4. Patients who underwent major surgery, open biopsy or significant traumatic injury within 4 weeks prior to the first dose of study drug.
5. Serious non-healing wound/ulcer/bone fracture.
6. ≥ grade 3 bleeding episodes within 6 months prior to first dose of study treatment, or currently ≥ grade 2 hemorrhage, with high bleeding risks (such as coagulation disorders, tracheobronchial infiltration with significant bleeding, active gastrointestinal ulcer and esophageal varices)
7. Active hemoptysis or more than 0.5 teaspoon (2.5 mL) of hemoptysis per day within 2 months before first dose of study treatment
8. Subjects with antiplatelet agents treatment (low-dose aspirin ≤100 mg/day is permitted).
9. Current or previous severe retinopathy who, in the judgment of the Investigator or specialist, are not suitable for enrollment
10. Significant cardiovascular impairment, including but not limited to:

    1. Serious arrhythmia or cardiac conduct abnormality, such as degree II-III atrioventricular block or ventricular arrhythmia needs to be treated.
    2. QTcF interval extension (by the Fridericia formula): male >450 ms, female >480 ms
    3. Acute coronary syndrome, stroke, deep vein thrombosis, pulmonary- thromboembolism, arterial thrombosis, congestive heart failure, aortic dissection etc.
    4. New York Heart Association Class ≥ II
    5. Uncontrolled hypertension, as defined by a sustained blood pressure (BP) > 140/90 mmHg.
11. Known brain metastasis unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and with a stable dose of corticosteroid treatment before first dose of study treatment.
12. Interstitial lung disease or radiation pneumonia in need of glucocorticoids intervention
13. Subjects with malignant tumors in the last 5 years (not including non-melanoma skin cancer, breast cancer or cervical cancer in situ, and Non-Muscle-invasive bladder cancer have been cured)
14. Receiving chronic concomitant treatment of strong CYP3A4 inducers, CYP3A4 inhibitors or CYP3A4 substrate with a narrow therapeutic window within 2 weeks prior to study drug administration,
15. Prior treatment of BRAF inhibitors.
16. Has not recovered from toxicities caused by prior therapy to CTCAE ≤Grade 1 (except for ≤Grade 2 peripheral neuropathy, alopecia, and other events judged tolerable by the Investigator and without safety risks).
17. HIV antibodies or Treponema pallidum antibodies positive, active hepatitis B (HBV-DNA≤ 2×ULN allowed to enroll), hepatitis C virus (HCV) antibody-positive and HCV-RNA- positive, or other active hepatitis, clinically significant moderate-to-severe cirrhosis. Prophylactic antiviral therapy other than interferon are allowed.
18. Acute bacterial, viral or fungal infections (any infection requiring systemic treatment)
19. Females who are pregnant or breastfeeding.
20. Drug or alcohol dependents.
21. Significant disorder of neurology or mental disease or poorly compliance.
22. Subjects with oral administration impossible, or in the conditions of malabsorption as determined by the investigator, such as dysphagia and intestinal obstruction, etc..
23. Uncontrolled pleural effusion, pericardial effusion, abdominal effusion requiring frequent drainage or medical intervention (clinically significant recurrence requiring additional intervention within 2 weeks after intervention, excluding exudate cytology) before first dose of study treatment.
24. Any history of other serious systemic diseases, or any other reason that might interfere with participation in trial or interfere with interpretation of trial results, in the judgement of the Investigator, that are not qualified to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  ORR is defined as the proportion of patients who have had a PR or CR as assessed by the RECIST 1.1. (CR: Complete Response, Disappearance of all target lesions, PR: Partial Response, >=30% decrease in the sum of the longest diameters of target lesions). Overall Response (OR) = CR + PR

SECONDARY OUTCOMES:
The number and frequency of treatment-related adverse events (AEs) and treatment related serious adverse events (SAEs) | Up to 24 months
  AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
PFS | Up to 24 months
  Progression-Free Survival (PFS) per RECIST 1.1
PFS6m | up to 24 months
  PFS6m per RECIST 1.1
DCR | up to 24 months
  Disease Control Rate (DCR) per RECIST 1.1
DOR | up to 24 months
  Duration of Response (DOR) per RECIST 1.1
OS | up to 24 months
  Overall Survival (OS) per RECIST 1.1
Thyroglobulin (Tg) | Up to 24 months
  Correlation analysis between Tg and efficacy of ST-1898
Thyroglobulin Antibody (TgAb) | Up to 24 months
  Correlation analysis between TgAb and efficacy of ST-1898
Pharmacokinetic (PK) Parameter: Tmax | On Day 1 from Cycle 1 to Cycle 4 (21 days per cycle), up to 12 weeks
  Time to Peak Plasma Concentration.
Pharmacokinetic (PK) Parameter: T1/2 | On Day 1 from Cycle 1 to Cycle 4 (21 days per cycle), up to 12 weeks
  Terminal Elimination Half-life.
Pharmacokinetic (PK) Parameter: Cmax | On Day 1 from Cycle 1 to Cycle 4 (21 days per cycle), up to 12 weeks
  Maximum Plasma Concentration.
Pharmacokinetic (PK) Parameter: AUC | On Day 1 from Cycle 1 to Cycle 4 (21 days per cycle), up to 12 weeks
  Area Under the Curve of ST-1898 plasma concentration-time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, Ph D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No